CLINICAL TRIAL: NCT02157454
Title: Randomized Controlled Trial to Evaluate the Effect of a Website Offering Individual Patient's Experiences on Patient Competence of Colorectal Cancer Patients
Brief Title: Effect of a Website Offering Individual Patients' Experiences for Cancer Patients
Acronym: DIPExRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berlin School of Public Health (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Principal Investigator, Christine Holmberg, Dr., MPH, Berlin School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NKP-332-041
Record Dates: First submitted 2014-05-27; First posted 2014-06-06 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Website access (Experimental): Two-week access to the colorectal cancer module of the website www.krankheitserfahrungen.de
  Interventions: Other: Website access
- Control (No Intervention): Participants who are randomized to the control group don't have access to the website until they have finished the last questionnaire at 6 weeks follow up.

INTERVENTIONS:
Other: Website access — Access to the colorectal cancer module of the website www.krankheitserfahrungen.de which provides free, reliable information about health issues by sharing people's real-life experiences
  Arms: Website access

SUMMARY:
Being diagnosed with cancer confronts patients with a severe disease and they need to learn to deal with a range of new challenges. In order to support patients in the coping process, the website www.krankheitserfahrungen.de provides patients free, reliable information about health issues by sharing peoples' real-life experiences. In our project, the investigators developed a new module on the website for patients with colorectal cancer.

The objective of our study is to evaluate if access to the new colorectal cancer module on the website www.krankheitserfahrungen.de increases patient's competence.

The investigators will conduct a two-arm randomized controlled trial. Patients affected by colorectal cancer will be randomized into an intervention and a control group: the intervention group will have access for two weeks to the website www.krankheitserfahrungen.de (colorectal cancer module) with cancer patients´ experiences. Patients in the control group will not receive any intervention but will have access to the website for two weeks after completing the study.

Patient competence is measured by the self-efficacy component of the German short form of the Cancer Behavior Inventory via an online questionnaire at baseline and after two weeks. A second follow-up assessment will be implemented six weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colorectal cancer within the last 3 years or with metastases or relapse after colorectal cancer
* having access to internet

Exclusion Criteria:

* Patients diagnosed with colorectal cancer more than 3 years ago and without metastases or relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Self-efficacy for coping with cancer (measured by the German short form of the Cancer Behavior Inventory) | after 2 weeks

SECONDARY OUTCOMES:
Change in self-efficacy for coping with cancer (measured by the German short form of the Cancer Behavior Inventory) | At baseline and after 2 weeks
Change in self-efficacy for coping with cancer (measured by the German short form of the Cancer Behavior Inventory) | At baseline and after 6 weeks
Patient competence (assessed by a self-rating measure of patient competence in oncology in validation process) | After 2 weeks
Patient competence (assessed by a self-rating measure of patient competence in oncology in validation process) | After 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Berlin School of Public Health, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Giesler JM, Keller B, Repke T, Leonhart R, Weis J, Muckelbauer R, Rieckmann N, Muller-Nordhorn J, Lucius-Hoene G, Holmberg C. Effect of a Website That Presents Patients' Experiences on Self-Efficacy and Patient Competence of Colorectal Cancer Patients: Web-Based Randomized Controlled Trial. J Med Internet Res. 2017 Oct 13;19(10):e334. doi: 10.2196/jmir.7639. PMID 29030329